CLINICAL TRIAL: NCT04386954
Title: To Study Patency Rates and Outcomes of Renal Access Arteriovenous Fistulas for Hemodialysis in Patients With Chronic Renal Failure
Brief Title: Outcomes of Renal Access Arteriovenous Fistulas for Hemodialysis in Patients With Chronic Renal Failure
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Anil Sharma, Consultant Renal transplant and urology, Principal Investigator, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBSIndiag
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: End Stage Renal Disease
Keywords: Arteriovenous Fistula, dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: observational study — observation study

SUMMARY:
End stage renal disease cases has increased significantly in the last decade. There are various treatment modalities which are available for the ESRD patients. Treatment options includes haemodialysis, peritoneal dialysis and renal transplant. Renal transplant is considered as the best treatment for these patients. However, in developing countries like india feasibility of renal transplant is questionable due to the limited donors and logistic reasons. Therefore haemodialysis remains the most popular modality of treatment for such patients. Creation of vascular access is a necessary maneuver for hemodialysis but creation and maintenance of a well-functioning vascular access remains the most challenging problems for hemodialysis therapy There are various other reasons for the non maturation of arteriovenous fistula and these include increased age, diabetes mellitus, hypertension, smoking, coronary artery disease, obesity, decreased diameter of the cephalic vein and radial artery, atherosclerosis, and surgeon factor. As per our literature search , these factors has not been well studied in Indian population. Hence the aim of the present study is to identify the various risk factors for the primary failure of forearm and wrist arteriovenous fistulas for hemodialysis in patients with chronic renal failure in Indian population

DETAILED DESCRIPTION:
Pre-operatively all patients were advised soft ball arm exercise. Patients were instructed not to use the concerned arm for blood sampling. The morning dose of antihypertensive was skipped if the patient mean arterial blood pressure was less than 100 mm Hg. Modified Allens test was done pre operative to check for the patency of the palmar arch. Preoperative Doppler of the concerned limb was done one day prior to the procedure by the consultant radiologist. The ulnar artery, radial artery, and cephalic vein diameter were measured at the wrist and the forearm. They were imaged in both transverse and sagittal planes at the levels of venous stenosis or thrombosis and a venogram was considered. On the day of surgery, patient were advised to take light breakfast in the morning prior to the procedure. Patient were shifted inside the operation theatre and all American society anaesthesiologist standard monitors were attached. This included pulse oxymeter, non invasive blood pressure and electrocardiogram. Patients lie supine on the operating table and the arm selected for fistula creation was abducted to an angle of 90 degree and kept on an arm rest.

Under all aseptic precaution 10 ml of local anaesthetic agent (5ml 2% Lidocaine + 5 ml Normal saline) was injected just proximal to wrist joint. After waiting for 5 minutes and confirmimg its effect, a 2 cm skin incision was made in between the radial artery and cephalic vein in the distal forearm. First of all, cephalic vein was dissected free from the surrounding structures. The S shaped retractors were used for the proper exposure. All vein tributaries were ligated with 4-0 silk. Vein at the distal end of the incision was ligated and divided. A 20 G cannula was inserted and 10 ml of heparinized saline (1 unit ml-1) was injected into the cephalic vein. After this a 5 F infant feeding tube was inserted into the vein and another 10 ml of heparinised saline was injected. Radial artery is then identified and mobilized from the surrounding structures. Around one and half cm of radial artery is exposed. Bull dog clamps were applied both proximally and distally to occlude the blood flow. Then using 11 number scalpel blade an arteriotomy of approximately 1 cm was done. Similarly veinotomy of around 1.3 cm was done for cephalic vein using the potts scissor. Then end to side anastomosis was done using continuous 7-0 prolene sutures. Posterior wall was done first, followed by the anterior wall. After completing the procedure and achieving complete haemostatsis, fistula was palpated for the presence of immediate thrill. Tablet amoxicillin 500 mg with clavulanic acid 125 mg was given to all patients for 5 days and after each dialysis. Soft ball arm exercise was also advised till the fistula matures. Immediate surgical complications were noted.

ELIGIBILITY:
Inclusion Criteria:

* all patients who present to the institute for primary renal vascular access for hemodialysis

Exclusion Criteria:

* patients with previous failed attempts for vascular access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of end stage renal disease
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-04-14 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
The correlation of cephalic vein and radial artery diameter with success of arteriovenous fistula. | 6 months
  The correlation of cephalic vein and radial artery diameter with success of arteriovenous fistula at 1 week, 1 month and 6 months.

SECONDARY OUTCOMES:
The correlation of age, sex, diabetes melitus and hypertension with success of arteriovenous fistula. | 6 months
  The correlation of age, sex, diabetes melitus and hypertension with success of arteriovenous fistula at 1 week, 1 month and 6 months.
Success rate of av fistula | 6 months
  Success rate of av fistula at 1 week, 1 month and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: anil sharma, mch, Principal Investigator — ilbs
Locations (1):
- Ilbs, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Swai J, Zhao X, Noube JR, Ming G. Systematic review and meta-analysis of clinical outcomes comparison between different initial dialysis modalities in end-stage renal disease patients due to lupus nephritis prior to renal transplantation. BMC Nephrol. 2020 May 1;21(1):156. doi: 10.1186/s12882-020-01811-y. PMID 32357924
- [Background] Haller MC, Kainz A, Baer H, Oberbauer R. Dialysis Vintage and Outcomes after Kidney Transplantation: A Retrospective Cohort Study. Clin J Am Soc Nephrol. 2017 Jan 6;12(1):122-130. doi: 10.2215/CJN.04120416. Epub 2016 Nov 28. PMID 27895135
- [Background] Siddiqui MA, Ashraff S, Santos D, Rush R, Carline T, Raza Z. Predictive parameters of arteriovenous fistula maturation in patients with end-stage renal disease. Kidney Res Clin Pract. 2018 Sep;37(3):277-286. doi: 10.23876/j.krcp.2018.37.3.277. Epub 2018 Sep 30. PMID 30254852
- [Result] Hall RK, Myers ER, Rosas SE, O'Hare AM, Colon-Emeric CS. Choice of Hemodialysis Access in Older Adults: A Cost-Effectiveness Analysis. Clin J Am Soc Nephrol. 2017 Jun 7;12(6):947-954. doi: 10.2215/CJN.11631116. Epub 2017 May 18. PMID 28522655
- [Result] Robbin ML, Greene T, Cheung AK, Allon M, Berceli SA, Kaufman JS, Allen M, Imrey PB, Radeva MK, Shiu YT, Umphrey HR, Young CJ; Hemodialysis Fistula Maturation Study Group. Arteriovenous Fistula Development in the First 6 Weeks after Creation. Radiology. 2016 May;279(2):620-9. doi: 10.1148/radiol.2015150385. Epub 2015 Dec 22. PMID 26694050
- [Result] Glass C, Johansson M, DiGragio W, Illig KA. A Meta-analysis of Preoperative Duplex Ultrasound Vessel Diameters for Successful Radiocephalic Fistula Placement. J Vasc Ultrasound. 2009 Jun 1;33(2):65-8.
- [Result] Hou G, Yan Y, Li G, Hou Y, Sun X, Yin N, Feng G. Preoperative cephalic vein diameter and diabetes do not limit the choice of wrist radio-cephalic arteriovenous fistula. J Vasc Access. 2020 May;21(3):366-371. doi: 10.1177/1129729819879320. Epub 2019 Oct 3. PMID 31580187
- [Result] Weale AR, Bevis P, Neary WD, Boyes S, Morgan JD, Lear PA, Mitchell DC. Radiocephalic and brachiocephalic arteriovenous fistula outcomes in the elderly. J Vasc Surg. 2008 Jan;47(1):144-50. doi: 10.1016/j.jvs.2007.09.046. PMID 18178467
- [Result] Misskey J, Faulds J, Sidhu R, Baxter K, Gagnon J, Hsiang Y. An age-based comparison of fistula location, patency, and maturation for elderly renal failure patients. J Vasc Surg. 2018 May;67(5):1491-1500. doi: 10.1016/j.jvs.2017.08.080. Epub 2017 Dec 8. PMID 29224945
- [Result] Dunn J, Herscu G, Woo K. Factors influencing maturation time of native arteriovenous fistulas. Ann Vasc Surg. 2015;29(4):704-7. doi: 10.1016/j.avsg.2014.11.026. Epub 2015 Feb 26. PMID 25728334